CLINICAL TRIAL: NCT01668056
Title: The Role of Controlling Follicular Wave Emergence to Synchronize Ovarian Stimulation for in Vitro Fertilization
Brief Title: Synchronization of Ovarian Stimulation for in Vitro Fertilization With Follicular Wave Emergence
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1099/09
Record Dates: First submitted 2012-08-06; First posted 2012-08-17 (Estimated); Last update posted 2013-09-10 (Estimated); Status verified 2013-09

CONDITIONS: Infertility
Keywords: in vitro fertilization; ovarian stimulation; follicular waves; luteal phase
MeSH Terms: conditions — Infertility | interventions — Ovulation Induction; Chorionic Gonadotropin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Control (Active Comparator): Patients will be stimulated according to the conventional flexible GnRH antagonist protocol for IVF. Alfa follitropin (150IU a day) will be started on the third day of the menstrual cycle. Treatment monitoring will be done with transvaginal ultrasound scans and serum determinations of estradiol and progesterone 5 days after the start of gonadotropins and every each day thereafter. Once the leading follicle reaches 13 mm in mean diameter 0,25mg of cetrorelix acetate will be administered daily. Once at least two follicles reach 18mm or more in mean diameter 250 micrograms of choriogonadotropin alfa will be administered and 36 hours latter patients will undergo follicle aspiration for IVF. Embryos will be cryopreserved (vitrification) on the third or fifth day of development. Two months after women will undergo uterine preparation for embryo transfer.
  Interventions: Other: Control
- Ovulation induction (Experimental): Patients will be monitored with daily transvaginal ultrasound scans from the tenth day of the menstrual cycle on. When the dominant follicle reaches a mean diameter of 16mm or more, patients will receive 250 micrograms of choriogonadotropin alfa subcutaneously. Daily transvaginal ultrasound scans will be done starting two days after the administration of the medication until a cohort of ovarian follicles between 4-6 mm is seen (follicular wave emergence). From this point on patients will undergo the same stimulation protocol as Controls, i.e., flexible GnRH antagonist protocol.
  Interventions: Drug: Ovulation induction with choriogonadotropin alfa
- Dominant follicle aspiration (Experimental): Patients will be monitored with daily transvaginal ultrasound scans from the tenth day of the menstrual cycle on. When the dominant follicle reaches a mean diameter of 16mm or more, patients will then undergo aspiration of the dominant and all follicles greater than 10mm in mean diameter. aspiration will be transvaginal ultrasound guided and under sedation, as for oocyte retrieval. Oocytes eventually obtained at this first aspiration will not be used for IVF. Daily transvaginal ultrasound scans will be done starting the day after the follicular aspiration until a cohort of follicles between 4-6 mm is seen (follicular wave emergence). From this point on patients will undergo the same stimulation protocol as Controls, i.e., flexible GnRH antagonist protocol.
  Interventions: Procedure: Aspiration of the dominant follicle

INTERVENTIONS:
Drug: Ovulation induction with choriogonadotropin alfa — Administration of 250 micrograms of choriogonadotropin alfa subcutaneously when the dominant follicle of a natural menstrual cycle reaches 16mm or more of mean diameter. Verify if this intervention is able to induce follicular wave emergence and synchronize the start of the flexible GnRH antagonist protocol of ovarian stimulation with the start of a follicular wave.
  Arms: Ovulation induction
Procedure: Aspiration of the dominant follicle — Aspiration of all follicles greater than 10mm in mean diameter when the dominant follicle of a natural menstrual cycle reaches 16mm or more of mean diameter. Aspiration will be guided by transvaginal ultrasound. Verify if this intervention is able to induce follicular wave emergence and synchronize the start of the flexible GnRH antagonist protocol of ovarian stimulation with the start of a follicular wave.
  Arms: Dominant follicle aspiration
Other: Control — Conventional flexible GnRH antagonist protocol of ovarian stimulation for in vitro fertilization, with gonadotropin star at the third day of a natural menstrual cycle.
  Arms: Control

SUMMARY:
Ovarian stimulation is an important phase of in vitro fertilization (IVF) treatments. The harvest of a larger number of viable eggs per cycle compensate eventual laboratory difficulties and allow for the selection of embryos with higher implantation potential. In the current protocols, based on the most prevailing theory of ovarian follicular development, stimulation drugs are usually started on the second or third day after the beginning of menses. The follicular phase of the menstrual cycle is believed to be the only favorable moment for follicular development.

In the early 2000's a new model of human ovarian follicular development (follicular waves) has been proposed based on frequent transvaginal ultrasound observations between two ovulations. It has been shown that ovarian antral follicles develop in synchronous groups, two to three times in a cycle. In fact the follicular wave phenomenon has been initially described in the 80's on domestic animals, like the mare and the cow. Moreover, studies in these animals have shown that synchronizing the start of the ovarian stimulation drugs with the beginning of a follicular wave yields better results for assisted reproductive treatments. Consequently in ovarian stimulation protocols for animal assisted reproduction it is important to control the initiation of a follicular wave.

Current protocols of ovarian stimulation for IVF in women do not consider the start of a follicular wave to begin drug administration. Therefore the purpose of this study is to evaluate two methods to control the emergence of a follicular wave (ovulation induction and dominant follicle aspiration) and to investigate the effects of synchronizing ovarian stimulation for IVF with follicular wave emergence in women compared to one of the current stimulation protocols (flexible GnRH protocol).

ELIGIBILITY:
Inclusion Criteria:

* age < 35 years old
* body mass index: 19-30 kg/m2
* tubal or male factor infertility with indication of in vitro fertilization
* antral follicle count: 10-20
* normal uterus in transvaginal ultrasound scan
* FSH on the third day of the menstrual cycle below 12mUI/mL and estradiol below 80pg/mL
* male partner with at least 5 million motile sperm and 1% normal strict morphology on semen analyses

Exclusion Criteria:

* ovarian factor infertility
* non identification of one or both ovaries in the transvaginal ultrasound scan
* non treated endocrine disorders
* smoking habit
* endometriosis stage III -IV
* severe male factor infertility (less than one million sperm per mL of semen)

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2012-01; Primary Completion 2014-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Emergence of an ovarian follicular wave after dominant follicle aspiration or hCG administration | One year
  Evaluate if the aspiration of the dominant follicle is able to induce a follicular wave to emerge.
  Evaluate if administration of hCG is able to induce ovulation of a dominant follicle larger than 16mm and to induce a follicular wave to emerge.
  A follicular wave emergence is defined as an increase in the number of ovarian follicles smaller than 10mm seen at the transvaginal ultrasound scan after the interventions
Follicular growth pattern on ultrasound scan | One year
  Evaluate with periodic transvaginal ultrasound scan the size (mm), number and growth rate (mm/day) of ovarian follicles in each of the three groups

SECONDARY OUTCOMES:
Estradiol and progesterone levels during ovarian stimulation | One year
  Evaluate blood levels of estradiol (pg/mL) and progesterone (ng/mL) during ovarian stimulation in each of the three groups at each visit to evaluate the progress of treatment.
Number of mature oocytes retrieved | One year
  Evaluate the number of metaphase II oocytes retrieved in each of the three groups
Total dose of gonadotrophins used | One year
  Total dose of gonadotrophins (in international units) necessary to stimulate the ovaries (from the first day of stimulation until the last dose of recombinant FSH administered before the oocyte retrieval)
Fertilization rate | One year
  Number of embryos formed in relation with the number of oocytes inseminated
Pregnancy rate | One year
  Positive beta hCG determination on blood 10 days after embryo transfer

CONTACTS AND LOCATIONS:
Overall Officials: Edmund c Baracat, PhD, Study Chair — University of Sao Paulo Medical School; Paulo C Serafini, PhD, Study Director — University of Sao Paulo Medical School; Paulo HM Bianchi, MD, Principal Investigator — University of Sao Paulo Medical School
Locations (1):
- University of Sao Paulo General Hospital, São Paulo, São Paulo, Brazil

REFERENCES:
- [Background] Baerwald AR, Adams GP, Pierson RA. A new model for ovarian follicular development during the human menstrual cycle. Fertil Steril. 2003 Jul;80(1):116-22. doi: 10.1016/s0015-0282(03)00544-2. PMID 12849812
- [Background] Baerwald AR, Adams GP, Pierson RA. Characterization of ovarian follicular wave dynamics in women. Biol Reprod. 2003 Sep;69(3):1023-31. doi: 10.1095/biolreprod.103.017772. Epub 2003 May 14. PMID 12748128
- [Background] Baerwald AR, Adams GP, Pierson RA. Ovarian antral folliculogenesis during the human menstrual cycle: a review. Hum Reprod Update. 2012 Jan-Feb;18(1):73-91. doi: 10.1093/humupd/dmr039. Epub 2011 Nov 8. PMID 22068695
- [Background] Adams GP, Singh J, Baerwald AR. Large animal models for the study of ovarian follicular dynamics in women. Theriogenology. 2012 Nov;78(8):1733-48. doi: 10.1016/j.theriogenology.2012.04.010. Epub 2012 May 22. PMID 22626769
- [Background] de Mello Bianchi PH, Serafini P, Monteiro da Rocha A, Assad Hassun P, Alves da Motta EL, Sampaio Baruselli P, Chada Baracat E. Review: follicular waves in the human ovary: a new physiological paradigm for novel ovarian stimulation protocols. Reprod Sci. 2010 Dec;17(12):1067-76. doi: 10.1177/1933719110366483. Epub 2010 May 3. PMID 20439948
- [Derived] Bianchi PH, Viera LM, Gouveia GR, Rocha AM, Baruselli PS, Baracat EC, Serafini PC. Study of two strategies to induce follicular wave emergence for assisted reproductive treatments (ART)-a preliminary trial. J Assist Reprod Genet. 2015 Apr;32(4):543-9. doi: 10.1007/s10815-015-0432-3. Epub 2015 Feb 21. PMID 25701140